CLINICAL TRIAL: NCT03522701
Title: Effects of Self-help Versus Group Cognitive Behavioural Therapy for Insomnia in Youth: a Randomised Controlled Trial
Brief Title: Effects of Self-help Versus Group Cognitive Behavioural Therapy for Insomnia in Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1710023
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Insomnia
Keywords: Adolescents; Youth; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A randomised, assessor-blind, parallel group controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group CBTI (Experimental): Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I) The intervention will consist of 8 weekly group sessions (90-min, 5-8 adolescents in each group) of CBT-I delivered within a 10-week window. The treatment components in the CBT-I aim to address the behavioural, cognitive and physiological perpetuating factor of insomnia and include: psycho-education about sleep and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Interventions: Behavioral: CBTI
- Email-delivered CBTI (Active Comparator): The email delivered self-guided CBT-I consists of 8 weekly learning sessions. Participants will receive an email embedded with session materials each week.
  Interventions: Behavioral: CBTI
- Waiting-list control (No Intervention): Participants will not receive any active treatment.

INTERVENTIONS:
Behavioral: CBTI — Refer to the arm description
  Arms: Email-delivered CBTI; Group CBTI

SUMMARY:
Insomnia is the most prevalent sleep problem in both the general and clinical populations. Insomnia symptoms, presented as the problems initiating sleep or maintaining sleep, have been reported in association with adverse outcomes in adolescents, including an increased risk of developing depression, anxiety, interpersonal problems, somatic health problems, self-harm and suicidal ideation. Moreover, adolescent insomnia has been found to predict the development of mental health problems in young adulthood.

Currently there is no medication specifically approved for use as hypnotics in children under age 18 by the US Food and Drug Administration (FDA). Although cognitive behavioural therapy for insomnia (CBT-I) has been regarded as the first-line treatment for insomnia in adults, there exists limited evidence for the efficacy of CBT-I among adolescents and young adults. Given the high prevalence and profound consequences of insomnia among youth, further research on the short-term and long-term effects of CBT-I for adolescents is warranted. To address the limitations of the existing literature, this randomised controlled trial aims to examine whether face-to-face (group-based CBT-I) versus self-help insomnia treatment benefit adolescents with insomnia, for improving sleep and other clinical and daytime symptoms as well as overall functional improvement in both the short and long term.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 12-24 years old (according to World Health Organization's defined age range for youth);
2. Written informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18);
3. Being able to comply with the study protocol;
4. Having a diagnosis of insomnia disorder, with a score on Insomnia Severity Index (ISI) >= 9 (suggested cut-off for adolescents)

Exclusion Criteria:

1. A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities;
2. Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. eczema, gastro-oesophageal reflux disease);
3. Having a clinically diagnosed sleep disorder that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome, as ascertained by the Diagnostic Interview for Sleep Patterns and Disorders (DISP);
4. Concurrent, regular use of medications(s) known to affect sleep continuity and quality (e.g. hypnotics, steroids);
5. In the opinion of the research clinician, having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt);
6. Having been enrolled in any other clinical trial investigational products within one month at the entry of the study;
7. Initiation of or change in antidepressant medication within past 2 months;
8. Having been or is currently receiving any structured psychotherapy;
9. With hearing or speech deficit;
10. Night shift worker.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of insomnia symptoms | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Insomnia Severity Index (ISI) is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change of sleep quality | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change of sleep diary measure (time in bed, TIB) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups]
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change of sleep diary measure (total sleep time, TST) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change of sleep diary measure (sleep onset latency, SOL) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups]
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins
Change of sleep diary measure (wake after sleep onset, WASO) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins
Change of sleep diary measure (sleep efficiency, SE) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change of objective sleep measure (time in bed, TIB) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours
Change of objective sleep measure (total sleep time, TST) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours
Change of objective sleep measure (sleep onset latency, SOL) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins
Change of objective sleep measure (wake after sleep onset, WASO) | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins
Change of daytime sleepiness | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change of daytime fatigue | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change of quality of life | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of suicidal ideation | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Depressive Symptom Inventory Suicidality Subscale (DSI-SS) is a 4-item self-rated scale measuring suicidal ideation. Possible total scores range from 0 to 12, with higher scores indicating higher suicidal ideation.
Change of self-report mood symptoms | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Hospital Anxiety and Depression Scale (HADS) is a self-assessed scale for detecting states of depression and anxiety. The depression subscale range in scores from 0 to 21, with higher scores indicating severer states of depression. Similarly, the anxiety subscale range in scores from 0-21 with higher scores indicating severer states of anxiety. No additional computation will be made with the two subscores
Change of dysfunctional beliefs and attitudes about sleep | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change of sleep hygiene and practice | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Sleep Hygiene Practice Scale (SHPS) is a 30-item self-rated scale measuring sleep hygiene behaviors, ranging in total scores from 30 to 180, with higher scores indicating lower levels of sleep hygiene.
Change of pre-sleep arousal | Baseline, post-treatment (week 8/at the conclusion of last session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups]
  Pre-Sleep Arousal Scale is a 16-item self-rated scale measuring pre-sleep arousal. There are two subscales on the cognitive and somatic manifestations of arousal, with eight items in each subscale (possibly scored from 8 to 40). In both cases, a higher score indicates higher pre-sleep arousal.
Change of depressive symptoms (assessor-rated) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Hamilton Depression Rating Scale (HAM-D): 17 item for assessing depression
Change of overall severity of clinical symptoms | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Clinical Global Impression (CGI) Scale is a clinician-rated scale, comprised of two one-item subscales: Severity of Illness (CGI-S) subscale evaluating the severity of the illness, and Clinical Global Improvement Scale (CGI-I) evaluating change from the initiation of treatment. In both cases, the score is given on a seven-point scale, with higher values indicating higher severity of illness and larger improvement respectively.
Change of objective cognitive performance (visual attention & task switching) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Trail Making Test for assessing visual attention and task switching. In Trail Making Test, longer reaction time indicates lower level of attention.
Change of objective cognitive performance (inhibitory ability) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Go/No-go Task for assessing inhibitory ability. In Go/No-go Task, a higher error rate indicates lower inhibition control.
Change of objective cognitive performance (working memory by digit span) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Digit Span Task for assessing working memory capacity. In Digit Span Task, a higher number of recalled digits indicates better working memory.
Change of objective cognitive performance (working memory by N-Back) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  N-back Task for assessing working memory capacity and manipulation. In N-back Task, a d prime score will be calculated based on the signal detection theory, where a higher score indicates better working memory performance.
Change of objective cognitive performance (episodic memory) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Chinese Auditory Verbal Learning Task for assessing episodic memory, where a higher number of recalled words indicates better episodic memory performance.
Change of objective cognitive performance (problem solving) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Wisconsin Card Sorting Test for assessing problem solving. In Wisconsin Card Sorting Test, lower executive functioning is indicated by a higher percentage of persistent errors and a higher number of trials taken to complete the first category.
Change of sleep related attention bias | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Sleep-related Dot-Probe Task for assessing sleep-related attention bias. In the Sleep-related Dot-probe Task, a higher attention bias score indicates higher vigilance towards sleep-related stimuli.
Change of risk-taking & decision making | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Balloon Analogue Risk Task for assessing risk-taking and decision-making. In Balloon Analogue Risk Task, a score will be calculated by averaging the number of pumps on unexploded blue balloons, where a higher score indicates more risk-taking and impulsive propensities.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, PhD, DClinPsy, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No